CLINICAL TRIAL: NCT02469831
Title: The Impact of Deep Versus Moderate Neuromuscular Block on Respiratory System Mechanics and Metabolic Changes During Laparoscopic Cholecystectomy a Double-Blind Randomized Clinical Trial.
Brief Title: Respiratory Mechanics and Metabolic Changes During Low Pressure Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, khaled salah mohamed, lecturer of anaesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: low pressure lap chole.
Record Dates: First submitted 2015-05-24; First posted 2015-06-12 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- group D (Active Comparator): deep neuromuscular block by rocuronium defined :post tetanic (PTC) >1 but no response to a train of four (TOF) stimulation.
  Interventions: Drug: Rocuronium
- group I (Active Comparator): intermediate neuromuscular block by rocuronium defined as TOF count of 1-3.
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium

SUMMARY:
The investigators aim to investigate the differences between deep continuous muscle relaxation and moderate blockade during low-pressure (8 mmHg) laparoscopic cholecystectomy in respect to metabolic changes and respiratory mechanics.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years
* undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* previous surgeries,
* a history of venous or arterial diseases,
* BMI (≥30 kg/m2),
* Allergy to rocuronium.
* Significant liver dysfunction.
* Significant renal dysfunction (S-creatinine > 200 umol/l).
* Neuromuscular disease that might impair neuromuscular blockade
* Pregnant or breastfeeding.
* Indication for rapid sequence induction.
* Inability to informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
respiratory mechanics (Dynamic compliance) | intraoperative
  Dynamic compliance

SECONDARY OUTCOMES:
surgeon satisfaction (scale from 1 to 5) | intraoperative
  scale from 1 to 5
postoperative pain (VAS score) | postoperative for 6 hours
  VAS score
postoperative nausea and vomiting | postoperative for 6 hours
completion of surgical procedure | intraoperative
  yes or no
metabolic changes (blood lactate) | intraoperative
  blood lactate

CONTACTS AND LOCATIONS:
Overall Officials: Osama ibraheim, MD, Study Chair — Assiut University; MOSTAFA ABBAS, MD, Study Chair — Assiut University; AHMED TAHA, MD, Study Chair — Assiut University
Locations (1):
- Al Rajhy liver hospital, Asyut, Asyut Governorate, Egypt